CLINICAL TRIAL: NCT01004718
Title: A Pilot Study to Assess the Feasibility of Detection and Quantification of Differences in Hodgkin Lymphoma and Diffuse Large B-cell Lymphoma Using FDG-PET/CT Imaging
Brief Title: Detection and Quant of Differences in Hodgkin Lymphoma and Diffuse Large B-cell Lymphoma Using Positron Emission Tomography/Computed Tomography (PET/CT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 21408; NCI-2009-01348
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Fluorodeoxyglucose F18; Fluorine-18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fludeoxyglucose F18 (FDG) PET/CT scans (Experimental): Patients undergo fludeoxyglucose F18 (FDG) positron emission tomography/computed tomography scans and 180 minutes after FDG administration.
  Interventions: Radiation: Fludeoxyglucose F18; Procedure: Computed Tomography; Procedure: Positron emission tomography

INTERVENTIONS:
Radiation: Fludeoxyglucose F18 — Undergo FDG PET/CT scans
  Other Names: 18FDG, FDG, Fluorine-18, 2 Fluoro-2-deoxy-D-Glucose, Fludeoxyglucose F18
Procedure: Computed Tomography — Undergo FDG PET/CT scans
  Other Names: tomography, computed
Procedure: Positron emission tomography — Undergo FDG PET/CT scans
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed

SUMMARY:
RATIONALE: Imaging procedures, such as positron emission tomography or computed tomography, may help in detecting differences between Hodgkin lymphoma or diffuse large B-cell lymphoma cancer cells. PURPOSE: This clinical trial is studying positron emission tomogaphy and computed tomography in determining differences in Hodgkin lymphoma and diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Assess the feasibility of detection and quantification of differences in the temporal and spatial distribution of FDG uptake between lesions of HL and DLBCL.

OUTLINE:

Patients undergo fludeoxyglucose F18 (FDG) positron emission tomography/computed tomography scans 60 and 180 minutes after FDG administration.

After completion of study, patients are followed for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a pathologically-proven diagnosis of classic HL or DLBCL with measurable disease by any imaging technique or physical examination.

Exclusion Criteria:

* Pregnant or nursing,
* Uncontrolled diabetes mellitus,
* Active infection,
* Inability to give informed consent or to comply with all study procedures,
* Subjects may be excluded at the discretion of the principal investigator or study team members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05; Primary Completion 2013-07 (Actual); Study Completion 2014-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fludeoxyglucose F18 (FDG) PET/CT Scans
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fludeoxyglucose F18 (FDG) PET/CT Scans
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 47 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Maximum Lesional FDG Uptake From 60 to 180 Minutes After FDG Administration
Description: Lesional fluorodeoxyglucose (FDG) uptake is measured by standardized uptake value (SUV). The study compared the percentage of change in maximum SUV over 2 hours (first measure was 60 minutes post-administration and second timepoint was 180 minutes post-administration).
Time Frame: 2 hours (between 60 minutes post-administration and 180 minutes post-administration)
Measure: Mean (Standard Deviation); unit: percentage of change in maximum SUV
Groups:
- Diffuse Large B-cell Lymphoma; Hodgkin's Lymphoma: Patients undergo fludeoxyglucose F18 (FDG) positron emission tomography/computed tomography scans and 180 minutes after FDG administration.
Arm/Group | Diffuse Large B-cell Lymphoma | Hodgkin's Lymphoma
Number analyzed (Participants) | 5 | 5
percentage of change in maximum SUV | 36.2 (12.4) | 32 (11.6)

ADVERSE EVENTS:
Arm/Group | Fludeoxyglucose F18 (FDG) PET/CT Scans
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes